CLINICAL TRIAL: NCT06857370
Title: Inter-lot Consistency Clinical Trial of Adsorbed Cell-free DTP (Three-component) Combined Vaccine
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTP-DTcP-003
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-02

CONDITIONS: Diphtheria, Tetanus and Acellular Pertussis
Keywords: Vaccine; Three Components; Immunogenicity; Safety; 2 months old
MeSH Terms: conditions — Diphtheria; Tetanus | interventions — Tetanus Toxoid; Vaccines, Combined

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental vaccine group A, 2 months old (Experimental): 3 doses of DTcP vaccine (0.5 ml) on Day 0and Month 2,4
  Interventions: Biological: Diphtheria, Tetanus and Acellular Pertussis (Three Components) Combined Vaccine, Adsorbed (DTcP Lot 1)
- Experimental vaccine group B, 2 months old (Experimental): 3 doses of DTcP vaccine (0.5 ml) on Day 0and Month 2,4
  Interventions: Biological: Diphtheria, Tetanus and Acellular Pertussis (Three Components) Combined Vaccine, Adsorbed (DTcP Lot 2)
- Experimental vaccine group C, 2 months old (Experimental): 3 doses of DTcP vaccine (0.5 ml) on Day 0and Month 2,4
  Interventions: Biological: Diphtheria, Tetanus and Acellular Pertussis (Three Components) Combined Vaccine, Adsorbed (DTcP Lot 3)

INTERVENTIONS:
Biological: Diphtheria, Tetanus and Acellular Pertussis (Three Components) Combined Vaccine, Adsorbed (DTcP Lot 1) — Three doses of basic immunization were completed at 2, 4 and 6 months of age
  Arms: Experimental vaccine group A, 2 months old
Biological: Diphtheria, Tetanus and Acellular Pertussis (Three Components) Combined Vaccine, Adsorbed (DTcP Lot 2) — Three doses of basic immunization were completed at 2, 4 and 6 months of age
  Arms: Experimental vaccine group B, 2 months old
Biological: Diphtheria, Tetanus and Acellular Pertussis (Three Components) Combined Vaccine, Adsorbed (DTcP Lot 3) — Three doses of basic immunization were completed at 2, 4 and 6 months of age
  Arms: Experimental vaccine group C, 2 months old

SUMMARY:
This is a randomized, blinded, peer-controlled study. There will be 3 treatment groups, screened subjects were randomized in a 1:1:1 ratio to receive three batches of the DTcP trial vaccine, and completed the primary immunization according to the procedure of one dose each at 2, 4, and 6 months of age.

ELIGIBILITY:
Inclusion Criteria:

* 2 months of age (60~89 days), willing to provide identification documents;
* The legal guardian or delegate has given informed consent, voluntarily signed the informed consent form, and can comply with the requirements of the clinical research protocol.

Exclusion Criteria:

First dose exclusion criteria

* Persons who have received a vaccine containing the DPT classified vaccine;
* Premature labor (delivery before 37th week of gestation), low birth weight 60 (birth weight <2500g);
* Those with abnormal labor and delivery, history of asphyxia rescue, history of neurological damage;
* Who have had one of the pertussis, diphtheria or tetanus diseases;
* Who have had household contact with an individual diagnosed with pertussis, diphtheria, or tetanus disease in the past 30 days;
* Have a history of allergy to vaccines or vaccine components and severe side reactions to vaccines, such as hives, dyspnea, angioneurotic edema, and other allergic reactions;
* Persons with a history of seizures, convulsions, convulsions, or cerebral palsy; or a history or family history of psychiatric illness; or other progressive neurologic disorders;
* Have been diagnosed with an immunodeficiency, Human Immunodeficiency Virus (HIV) infection, lymphoma, leukemia, Systemic Lupus Erythematosus (SLE), Juvenile Rheumatoid Arthritis ( Juvenile Rheumatoid Arthritis (JRA) or other autoimmune diseases;
* Any condition resulting in absence of spleen, defective spleen function;
* Known or suspected acute illness or severe chronic disease (including: severe respiratory disease, severe cardiovascular disease, liver or kidney disease, severe skin disease, malignancy, etc.); or in an acute exacerbation of a chronic disease;
* Physician-diagnosed coagulation abnormalities (e.g., coagulation factor deficiencies, coagulopathies, platelet abnormalities) or significant bruising or coagulation disorders;
* Immunosuppressive or modifying agents, cytotoxic consecutive therapy for more than 10 days (except inhaled and topical steroids) within 2 months prior to receiving the test vaccine;
* Received blood products (other than hepatitis B immune globulin) within 2 months prior to receiving the test vaccine;
* Participated or planning to participate in any other drug or vaccine clinical study;
* Has received an injectable live attenuated vaccine within 14 days or another vaccine within 7 days prior to receiving the test vaccine;
* Axillary temperature >37.3°C prior to vaccination;
* Any other factor that, in the investigator's judgment, makes the subject unsuitable for participation in a clinical trial.

Exclusion Criteria for Doses 2,3

* Persons who have had a severe allergic reaction following a previous dose of vaccine;
* Persons with serious adverse reactions causally related to the previous dose of vaccination;
* Those with a newly identified or newly occurring condition after the first dose of vaccination that does not meet the inclusion criteria for the first dose or meets the exclusion criteria for the first dose, as determined by the investigator for continued participation in the study;
* Other reasons for exclusion as determined by the investigator.

Ages: 60 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 780 (Actual)
Dates: Start 2025-03-23 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Geometric Mean Concentration (GMC) of serum anti-PT, FHA, PRN, DT, and TT antibodies in 2-month-old subjects with three different batches of the trial vaccine. | 30 days after vaccination

SECONDARY OUTCOMES:
Seroconversion rate of serum anti-PT, FHA, PRN, DT, and TT antibodies in 2-month-old subjects with three different batches of the trial vaccine. | 30 days after vaccination
Seropositivity rate of serum anti-PT, FHA, PRN, DT, and TT antibodies in 2-month-old subjects with three different batches of the trial vaccine | 30 days after vaccination
Incidence of solicited adverse reactions for each vaccine dose in 2-month-old subjects. | Within 30 minutes post-vaccination
Incidence of solicited adverse reactions for each vaccine dose in 2-month-old subjects. | Within 0-7 days
Incidence of unsolicited adverse reactions for each vaccine dose in 2-month-old subjects. | Within 0-30 days
Incidence of Serious Adverse Events (SAEs) in 2-month-old subjects. | From first vaccination to 30 days after the third dose

CONTACTS AND LOCATIONS:
Overall Officials: Yanxia Wang, Principal Investigator — Henan Center for Disease Control and Prevention
Locations (1):
- Changge Center for Disease Control and Prevention, Xuchang, Henan, China